CLINICAL TRIAL: NCT05559203
Title: A Realist Evaluation of the Feasibility of a Digital Music and Movement Intervention for Older People Living in Care Homes
Brief Title: danceSing Care Evaluation: Testing the Feasibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stirling (Other)
Responsible Party: Principal Investigator, Anna Whittaker, Principal Investigator, University of Stirling
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NICR 3735
Record Dates: First submitted 2022-09-08; First posted 2022-09-29 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Aged; Older Adults; Healthy Aging; Aging
Keywords: feasibility study; realist evaluation; care homes; clinical trial; physical activity; digital intervention; music and movement intervention; dance intervention
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Digital music and movement resources.
  Interventions: Behavioral: danceSing Care

INTERVENTIONS:
Behavioral: danceSing Care — The programme was a digital movement and music programme with resources from danceSing Care and consisted of three movement sessions and one music session each week, the recommended dose agreed between danceSing Care and the Advisory group, each lasting about 20 minutes. Also, the danceSing care resources were designed to suit older adults with physical and cognitive impairments (residents with mobility aids and/or dementia). Movement sessions included chair and standing fitness, which started with a warm-up and finished with stretching exercises. Sessions were managed and supervised by care home activity coordinators.

SUMMARY:
* The investigators wanted to find out if digital music and movement resources could be delivered in care homes. They rolled out a 12-week programme to 10 care homes and had 47 care home residents participate in the research.
* The investigators also wanted to find out under what circumstances the digital music and movement resources would be most effective for the health and wellbeing of the care home residents.
* A survey measuring the number of falls in the past three months, activities of daily living and health, psychosocial wellbeing (anxiety, depression, stress and loneliness), sleep satisfaction and frailty measures such as appetite and weight loss) was completed before and after the intervention. Also, interviews with residents and focus groups with staff were done after the intervention to find out how they felt about the programme.

DETAILED DESCRIPTION:
The specific research objectives were to evaluate the following topics:

1. Feasibility: was the activity implemented and/or delivered as planned? Were the resources suitable for this setting? Were adherence rates at an acceptable level?
2. Context: what is the role of the care homes in providing resources to the Activity Coordinators (ACs)? In what circumstances would the programme have worked most efficiently? What were the potential barriers for care homes or ACs to provide these resources?
3. Mechanism: what underlying mechanisms made the danceSing Care programme work (or not)? Was it the situational context or the programme context?
4. Outcome: What were the results? Were the outcomes adequate and realistic for this programme?
5. Moderators: were moderating factors responsible? By moderating factors, we are referring to contextual factors that are out of the program's control but may help or hinder the achievement of the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* residents in care homes ≥ 65 years,
* able to complete 12 weeks of a movement and music program,
* having the capacity to give informed consent.

Exclusion Criteria:

* currently taking part in any other clinical trial which could potentially have an impact upon or influence the findings of the current study,
* pre-existing conditions or concurrent diagnoses which would profoundly impact their capacity to undergo the intervention, even once adaptations have been made,
* inability to understand written/spoken English adequately to participate in the measures and intervention (e.g., due to cognitive or sensory impairment).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Whittaker, Principal Investigator — University of Stirling
Locations (1):
- Balhousie Care Group, Perth, United Kingdom

REFERENCES:
- [Result] Ofosu EF, De Nys L, Connelly J, Ryde GC, Whittaker AC. A realist evaluation of the feasibility of a randomised controlled trial of a digital music and movement intervention for older people living in care homes. BMC Geriatr. 2023 Mar 6;23(1):125. doi: 10.1186/s12877-023-03794-5. PMID 36879201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 did not meet eligibility criteria resulting in 47 participants enrolled across 10 care homes
Pre-assignment Details: did not meet age inclusion criterion
Units Other Than Participants: care homes
Groups:
- Single Arm Trial - Intervention Group n = 47 Participants Were Allocated the Intervention: Digital music and movement resources.
  danceSing Care: The programme was a digital movement and music programme with resources from danceSing Care (https://dancesingcare.uk/) and consisted of three movement sessions and one music session each week, the recommended dose agreed between danceSing Care and the Advisory group, each lasting about 20 minutes. Also, the danceSing care resources were designed to suit older adults with physical and cognitive impairments (residents with mobility aids and/or dementia). Movement sessions included chair and standing fitness, which started with a warm-up and finished with stretching exercises. Sessions were managed and supervised by care home activity coordinators.
Period: Overall Study
Arm/Group | Single Arm Trial - Intervention Group n = 47 Participants Were Allocated the Intervention
Started | 47; 10 care homes
Completed Intervention (The review considers the units to be care homes not participants, I have changed this so it matches the adherence outcomes, however, this brings us into difficulties for the other outcome analyses where it is across participants - people not homes) | 47; 10 care homes
Completed (completed follow-up data collection) | 33; 7 care homes
Not Completed | 14; 3 care homes
Not completed — Intervention not implemented at their care home due to insufficient staff | 14

BASELINE CHARACTERISTICS:
Population: older adults living in residential care homes - Scotland
Groups:
- Intervention Group n = 47 Allocated: Digital music and movement resources.
  danceSing Care: The programme was a digital movement and music programme with resources from danceSing Care (https://dancesingcare.uk/) and consisted of three movement sessions and one music session each week, the recommended dose agreed between danceSing Care and the Advisory group, each lasting about 20 minutes. Also, the danceSing care resources were designed to suit older adults with physical and cognitive impairments (residents with mobility aids and/or dementia). Movement sessions included chair and standing fitness, which started with a warm-up and finished with stretching exercises. Sessions were managed and supervised by care home activity coordinators.
Arm/Group | Intervention Group n = 47 Allocated
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 33

OUTCOME MEASURES:

1. Primary Outcome: Participants' Programme Adherence as % Sessions Attended Out of the Possible Maximum Number of Sessions Delivered Per Care Home Aggregated as % Across All Care Homes.
Description: The activity coordinators will fill in participants' adherence after each session. The completed files will be sent through to the investigators. Individual participants' adherence is calculated as the number of sessions they individually attended out of the possible number of sessions available to them in their care home. This is reported as the percentage of attended sessions per person per care home out of those delivered averaged per care home then aggregated across all care homes.
Time Frame: Will be evaluated after completion of the 12-week intervention period
Population: calculates the number of sessions attended on average out of the possible maximum number of sessions delivered
Measure: Count of Units; unit: Delivered Sessions
Units Other Than Participants: Delivered Sessions
Arm/Group | Intervention Group n = 47 Allocated
Number analyzed (Participants) | 33
Number analyzed (Delivered Sessions) | 193
Delivered Sessions | 116

2. Primary Outcome: Number of Sessions Delivered, Assessed by Attendance Files
Description: The activity coordinators will fill in participants' adherence after each session. The completed files will be sent through to the investigators.
Time Frame: Will be evaluated after completion after the completion of the 12-week intervention period
Population: Adherence across all carehomes allocated to the intervention, 7 delivered the intervention. Number of sessions delivered out of the recommended 48, then averaged across all 7 care homes.
Measure: Count of Units; unit: Delivered Sessions
Units Other Than Participants: Delivered Sessions
Arm/Group | Intervention Group n = 47 Allocated
Number analyzed (Participants) | 33
Number analyzed (Delivered Sessions) | 336
Delivered Sessions | 193

3. Primary Outcome: Acceptability of the Intervention Assessed by Focus Groups - Semi-structured Questions Covering Subjective Views on Enjoyment, Motivation, Duration, Content Etc.
Description: Investigators will conduct focus groups with the activity coordinators to assess acceptability of the intervention. Guide questions included:
  Did you enjoy using the danceSing Care online activities? Did you manage to take part in the 3+1 sessions a week? If not, why? Would you say duration of sessions was appropriate? Did you complete most of sessions or have to stop at any point? What did you like about the DSC activities? Was there anything you did not like? If you could change something about this programme to make it work effectively here, what would you change and why? Why did you take part? What made you continue to take part? What do you consider the outcomes of this program to have been for you? Would you like to carry on engaging in the DSC activities? Why/why not? Do you feel part of the DSC family/champions? Has engaging in the DSC activities brought you closer to other residents and staff?
Time Frame: 1 month after completion after the completion of the 12-week intervention period
Population: Five core themes emerged from 2 focus groups with 5 activity coordinators (care staff) across 2 focus groups. Exemplar quotes are given in the publication from this study.
Measure: Count of Units; unit: qualitative themes
Units Other Than Participants: qualitative themes
Arm/Group | Single Arm Trial - Intervention Group n = 47 Participants Were Allocated the Intervention
Number analyzed (Participants) | 5
Number analyzed (qualitative themes) | 5
qualitative themes
  Adherence - participation and class size | 1
  Delivery challenges with intervention | 1
  Intervention Effects | 1
  Modifications | 1
  Future Refinements | 1

4. Primary Outcome: Acceptability of the Intervention Assessed by Interviews - Semi-structured Questions Covering Subjective Views on Enjoyment, Motivation, Duration, Content Etc.
Description: Investigators will conduct focus groups/interviews with residents to assess acceptability of the intervention. Guide questions included:
  Did you enjoy using the danceSing Care online activities? Did you manage to take part in the 3+1 sessions a week? If not, why? Would you say duration of sessions was appropriate? Did you complete most of sessions or have to stop at any point? What did you like about the DSC activities? Was there anything you did not like? If you could change something about this programme to make it work effectively here, what would you change and why? Why did you take part? What made you continue to take part? What do you consider the outcomes of this program to have been for you? Would you like to carry on engaging in the DSC activities? Why/why not? Do you feel part of the DSC family/champions? Has engaging in the DSC activities brought you closer to other residents and staff?
Time Frame: 1 month after completion after the completion of the 12-week intervention period
Population: 4 residents in 4 semi-structured interviews. Exemplar quotes are in the publication of the study.
Measure: Count of Units; unit: qualitative themes
Units Other Than Participants: qualitative themes
Arm/Group | Intervention Group
Number analyzed (Participants) | 4
Number analyzed (qualitative themes) | 5
qualitative themes
  Adherence | 1
  Delivery challenges - Motivation and engagement | 1
  Modifications | 1
  Intervention Effects | 1
  Future Implementation | 1

5. Secondary Outcome: Change in Fear of Falling Between Baseline and Within One Month of Completing the Intervention Using the Falls Efficacy Scale - International (Short Form)(FES-I)
Description: It is a 16 item questionnaire, useful to the researchers and clinicians interested in fear of falling, with a score ranging from minimum 16 (no concern about falling) to maximum 64 (severe concern about falling).
Time Frame: Baseline and within 1 month of completion of the 12-week intervention period
Population: Only 18 participants retained capacity to continue to consent and capacity to complete follow-up measures. Outcomes are mean difference from baseline to post-intervention.
Measure: Mean (99% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group n = 47 Allocated
Number analyzed (Participants) | 18
units on a scale | -.556 [-4.199 to 3.088]
Statistical Analysis 1: Comparison: Intervention Group n = 47 Allocated; Feasibility study so no power calculation. N = 18 with baseline and follow-up data; Test type: Equivalence — 0.05 test of null hypothesis that there will be no significant change from baseline to post-intervention; p = .752, t-test, 2 sided; paired sample

6. Secondary Outcome: Change in Participant's Activities of Daily Living and Health-related Quality of Life From Baseline to Within One Month of the Completion of the Intervention Using The Dartmouth COOP Charts
Description: Change in participant's Activities of daily living and health-related quality of life from baseline to within one month of the completion of the intervention using The Dartmouth COOP which has 5-point Likert-type scaling, with descriptors and cartoon illustrations of levels 1 through 5. Rating of "1" = no impairment, "5" = most impaired.
Time Frame: Baseline and within 1 month of completion of the 12-week intervention period
Population: 18 with pre- and post-intervention data. Mean difference measure.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group n = 47 Allocated
Number analyzed (Participants) | 18
units on a scale | 1.167 [-.664 to 2.998]
Statistical Analysis 1: Comparison: Intervention Group n = 47 Allocated; Feasibility study so no power calculation. N = 18 with baseline and follow-up data; Test type: Equivalence — 0.05 test of null hypothesis that there will be no significant change from baseline to post-intervention; p = .197, t-test, 2 sided

7. Secondary Outcome: Change in Participant's Activities of Daily Living and Health-related Quality of Life From Baseline to Within One Month of Completing the Intervention Using EQ-5D-3L
Description: The EQ-5D-3L descriptive system comprises the following five questions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each question has a 3-point scale for rating it: no problems, some problems, and extreme problems (1-3). The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions are then combined to describe the patient's health state, with a higher TOTAL score describing a worse outcome. The range for total score is 5-15.
Time Frame: Baseline and within 1 month of completion of the 12-week intervention period
Population: 18 with pre- and post-intervention data. Mean difference measure between their TOTAL score at baseline and post-intervention.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group n = 47 Allocated
Number analyzed (Participants) | 18
units on a scale | .278 [-.714 to 1.270]
Statistical Analysis 1: Comparison: Intervention Group n = 47 Allocated; Test type: Equivalence — 0.05 test of null hypothesis that there will be no significant change from baseline to post-intervention; p = .562, t-test, 2 sided

8. Secondary Outcome: Change in Participant's Psychosocial Wellbeing From Baseline to Within One Month of Completing the Intervention Using the Hospital Anxiety and Depression Scale (HADS)
Description: The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression. No total score is reported. Anxiety and Depression sub-scale totals are calculated separately by summing responses to the applicable 7 items each. The range for each sub-scale is 0-21. A higher score indicates a worse outcome.
Time Frame: Baseline and within 1 month of completion of the 12-week intervention period
Population: 18 with pre- and post-intervention data. Mean difference measure. For anxiety and depression separately.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group n = 47 Allocated
Number analyzed (Participants) | 18
units on a scale
  Anxiety | 2.111 [.373 to 3.850]
  Depression | 3.0 [1.303 to 4.697]
Statistical Analysis 1: Comparison: Intervention Group n = 47 Allocated; Anxiety subscale; Test type: Equivalence — 0.05 test of null hypothesis that there will be no significant change from baseline to post-intervention; p = .020, t-test, 2 sided
Statistical Analysis 2: Comparison: Intervention Group n = 47 Allocated; Depression subscale; Test type: Equivalence — 0.05 test of null hypothesis that there will be no significant change from baseline to post-intervention; p = .002, t-test, 2 sided

9. Secondary Outcome: Change in Participant's Psychosocial Wellbeing From Baseline to Within One Month of Completing the Intervention Using the Perceived Stress Scale (PSS)
Description: Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Time Frame: Baseline and within 1 month of completion of the 12-week intervention period
Population: 18 with pre- and post-intervention data. Mean difference measure.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group n = 47 Allocated
Number analyzed (Participants) | 18
units on a scale | 4.167 [.318 to 8.016]
Statistical Analysis 1: Comparison: Intervention Group n = 47 Allocated; Test type: Equivalence — 0.05 test of null hypothesis that there will be no significant change from baseline to post-intervention; p = .036, t-test, 2 sided

10. Secondary Outcome: Change in Participant's Psychosocial Wellbeing From Baseline to Within One Month of Completing the Intervention Using the Brief UCLA Loneliness Scale (ULS-6)
Description: Using a 4-point rating scale (1= never; 4 = always), participants answer 6 questions, such as "How often do you feel left out?" and "How often do you feel part of a group of friends?". The Brief UCLA Loneliness scale is summed across items to give one total score. The range for total score is 6-24. A higher score indicates worse loneliness, i.e. a worse outcome.
Time Frame: Baseline and within 1 month of completion of the 12-week intervention period
Population: 18 with pre- and post-intervention data. Mean difference measure.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group n = 47 Allocated
Number analyzed (Participants) | 18
units on a scale | 1.667 [.067 to 3.267]
Statistical Analysis 1: Comparison: Intervention Group n = 47 Allocated; Test type: Equivalence — 0.05 test of null hypothesis that there will be no significant change from baseline to post-intervention; p = .042, t-test, 2 sided

11. Secondary Outcome: Change in Participant's Sleep Satisfaction From Baseline to Within One Month of Completing the Intervention Using the National Sleep Foundation's Sleep Satisfaction Tool (SST)
Description: 9-item questionnaire (scoring 1 not satisfied to 4 very satisfied) to assesses the general population's sleep satisfaction. The SST scale is summed across items to give one total score. The range for total score is 9-36.
Time Frame: Baseline and within 1 month of completion of the 12-week intervention period
Population: 18 with pre- and post-intervention data. Mean difference measure.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group n = 47 Allocated
Number analyzed (Participants) | 18
units on a scale | -6.667 [-9.174 to -4.159]
Statistical Analysis 1: Comparison: Intervention Group n = 47 Allocated; Test type: Equivalence — 0.05 test of null hypothesis that there will be no significant change from baseline to post-intervention; p < .001, t-test, 2 sided

12. Secondary Outcome: Change in Participant's Appetite From Baseline to Within One Month of Completing the Intervention Using the Simplified Nutritional Appetite Questionnaire (SNAQ)
Description: This is used for limited frailty testing, a self-assessment nutritional screening tool that predicts weight loss, scoring 1 (very poor) to 4 (very good) on appetite-related topics.
Time Frame: Baseline and within 1 month of completion of the 12-week intervention period
Population: 18 with pre- and post-intervention data. Mean difference measure.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group n = 47 Allocated
Number analyzed (Participants) | 18
units on a scale | .167 [-1.078 to 1.411]
Statistical Analysis 1: Comparison: Intervention Group n = 47 Allocated; Test type: Equivalence — 0.05 test of null hypothesis that there will be no significant change from baseline to post-intervention; p = .781, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: fall resulting in serious injury/hospitalisation
Arm/Group | Intervention Group n = 47 Allocated
All-Cause Mortality (participants affected / at risk) | 3/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/03/NCT05559203/Prot_SAP_001.pdf
  • Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT05559203/ICF_000.pdf